CLINICAL TRIAL: NCT01741935
Title: Is COPD Patient Mobility in Combination With Other Parameters a Sensitive Measure and Predictive Indicator for Early Detection of Exacerbations in COPD?
Brief Title: Continuous Monitoring of Patients With Chronic Obstructive Pulmonary Disease
Acronym: CTC-Actiwise
Status: Completed | Type: Observational
Sponsor: CareTelCom AB (Industry)
Collaborators: Boehringer Ingelheim (Industry); Region Skane (Other); Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: CTC002.1
Record Dates: First submitted 2012-11-22; First posted 2012-12-05 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An open, single group, single center Study to confirm CTC-Actiwise™ as a means to record and monitor the progression of a patient's COPD.

Chronic Obstructive Pulmonary Disease (COPD) affects growing patient groups. Current knowledge about the disease limits the investigators ability to cure or interfere with the progression of the disease. COPD is often characterized by exacerbating infections requiring emergency care.

The project aims to examine whether disease progression of COPD can be better controlled by continuously monitoring the patient's physical activity, along with the assessment of pulmonary symptoms and lung function. A key question is: can investigators find indicators that provides support for early intervention before severe symptoms arise.

The patient carries a smartphone that records physical activity real-time, daily lung function measures, lung disease related symptoms, and use of medication.

The experimental phase, the first part of the project, covers 25 COPD patients followed up to 12 weeks where the primary objective is to examine and verify both new investigational methodology and technology.

ELIGIBILITY:
Inclusion Criteria:

* Female or male 40 years of age and above
* Ability to use a smartphone and Bluetooth spirometer
* Subjects having COPD
* Ongoing treatment for a recent and not completely recovered COPD exacerbation

Exclusion Criteria:

* Dominating physical disability for other reasons or not related to COPD

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Improved real time physical activity | Patients are continuously monitored up to 12 weeks
  Improved health following an exacerbation is expected to be reflected by an increase in patient's physical activity performance recorded real time. The physical activity trend is compared with the trends in twice-daily recordings of symptom scores, use of rescue medication, and lung function. The correlation between the trends is measured.

SECONDARY OUTCOMES:
The correlation of physical activity to disease symptom scores, lung function, and use of medication | Patients are continuously monitored up to 12 weeks
  Improved health following an exacerbation is expected to be reflected by an increase in patient's physical activity performance recorded real time. The physical activity trend is compared with the trends in twice-daily recordings of symptom scores, use of rescue medication, and lung function. The correlation between the trends is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Leif Bjermer, Professor, Principal Investigator — Lund University
Locations (1):
- Department of Respiratory Medicine & Allergology, Skånes universitetssjukhus Lund, Lund, Sweden